CLINICAL TRIAL: NCT01560065
Title: Effect of Treatment With Myo-inositol on Human Semen Parameters in Patients Undergoing In Vitro Fertilization Cycles
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AGUNCO Obstetrics and Gynecology Centre (Other)
Responsible Party: Sponsor
Other Study IDs: MI_IVF
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-01

CONDITIONS: Sperm Quality; Oligoasthenospermia
MeSH Terms: interventions — Inositol; Folic Acid

ARMS (3):
- Normospermic patients (Other)
  Interventions: Dietary Supplement: myo-inositol + folic acid
- Oligoasthenospermic patients (Other)
  Interventions: Dietary Supplement: myo-inositol + folic acid
- Control (No Intervention)

INTERVENTIONS:
Dietary Supplement: myo-inositol + folic acid — 4000mg myo-inositol + 400 µg folic acid
  Arms: Normospermic patients
Dietary Supplement: myo-inositol + folic acid — 4000mg myo-inositol + 400 µg folic acid
  Arms: Oligoasthenospermic patients

SUMMARY:
Myo-Inositol (MI) is a precursors for the synthesis of phosphatidylinositol polyphosphates (PIPs). In male reproduction, it was shown that MI concentration in the seminiferous tubules is higher than in serum and it was increasing during the movement through the epididymis and the deferent duct. In the present study, the role of myo-inositol has been investigated as a possible antioxidant agent for the systemic treatment of male infertility and the improvement of the sperm's quality.

Samples of seminal fluid were obtained from two groups of patients undergoing to a IVF cycle: healthy subjects and subjects with oligoasthenospermia (OA, < 15 mil/ml). The collected samples were submitted to optic microscopy in order to evaluate semen's volume, spermatozoa's number and motility, during the initial semen analysis and after density gradient separation method; these parameters were evaluated before and after the administration of 4000mg/die of myo-inositol associated to 400 µg of folic acid for three months.

These values were compared with samples of seminal fluid of healthy patients undergoing to a IVF cycle for a female cause of infertility (control group).

ELIGIBILITY:
Inclusion Criteria:

* 3-5 days of sexual abstinence

Exclusion Criteria:

* systemic and endocrine diseases
* genital infections
* history of cryptorchidism or varicocele
* microorchidism
* hormonal treatment in the last six months
* alcohol intake, cigarette smoke and/or drug abuse

Ages: 18 Years to 40 Years | Sex: Male
Age Groups: Adult

PRIMARY OUTCOMES:
Semen volume
Spermatozoa count
Spermatozoa progressive motility
Number of spermatozoa after density gradient separation method

CONTACTS AND LOCATIONS:
Locations (1):
- University of Catania - Department of Surgery - Section of Obstetrics and Gynecology -Center of Physiopathology of Reproduction, Catania, Italy

REFERENCES:
- [Background] Colone M, Marelli G, Unfer V, Bozzuto G, Molinari A, Stringaro A. Inositol activity in oligoasthenoteratospermia--an in vitro study. Eur Rev Med Pharmacol Sci. 2010 Oct;14(10):891-6. PMID 21222378
- [Background] Hinton BT, White RW, Setchell BP. Concentrations of myo-inositol in the luminal fluid of the mammalian testis and epididymis. J Reprod Fertil. 1980 Mar;58(2):395-9. doi: 10.1530/jrf.0.0580395. PMID 7431272
- [Derived] de Ligny W, Smits RM, Mackenzie-Proctor R, Jordan V, Fleischer K, de Bruin JP, Showell MG. Antioxidants for male subfertility. Cochrane Database Syst Rev. 2022 May 4;5(5):CD007411. doi: 10.1002/14651858.CD007411.pub5. PMID 35506389